CLINICAL TRIAL: NCT00737412
Title: A Double-blind, Randomized, Placebo Controlled, Multicenter Study of the Efficacy of BIO-K+ CL1285® Prophylaxis in the Prevention of Traveler's Diarrhea in Adults.
Brief Title: Efficacy of BIO-K+ CL1285® Prophylaxis in the Prevention of Traveler's Diarrhea in Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bio-K Plus International Inc. (Industry)
Collaborators: ethica Clinical Research Inc. (Industry)
Responsible Party: Marcia T. Ruiz, Bio-K+ International Inc.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CL1285-TD-M02
Record Dates: First submitted 2008-08-15; First posted 2008-08-19 (Estimated); Last update posted 2010-01-21 (Estimated); Status verified 2010-01

CONDITIONS: Diarrhea
Keywords: Bio-K+CL1285; Probiotics; Traveler's Diarrhea; Lactobacillus Acidophilus; Lactobacillus Casei
MeSH Terms: conditions — Diarrhea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): The probiotic Bio-K+ CL1285 RX®
  Interventions: Other: Probiotic: Bio-K+ CL1285
- 2 (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Probiotic: Bio-K+ CL1285 — The probiotic Bio-K+ CL1285 RX®, a mixture of Lactobacillus acidophilus and Lactobacillus casei, contains over 50 billion living bacteria per administered dose.
  Other Names: Bio-K+ CL1285 RX®
  Arms: 1
Other: Placebo — Matching capsules devoid of microorganisms
  Arms: 2

SUMMARY:
The purpose of this study is to determine the efficacy of Bio-K+ CL1285 in reducing traveler's diarrhea.

DETAILED DESCRIPTION:
Determine efficacy of Bio-K+ CL1285 in reducing Traveler's Diarrhea by comparing the incidence of diarrhea in travelers during their stay abroad and upon their return to Canada following either Bio-K+ CL-1285 OR placebo prophylaxis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects over 18 years of age traveling to Mexico, Central America, South America and Caribbean Islands as direct destinations or on cruises to the same destinations.
* The trips last a minimum of 7 days and a maximum of 21 days.
* Women of child bearing capacity who are not pregnant at the moment of screening (pregnancy test done on-site) and agree to use an acceptable form of birth control for the duration of the study (e.g. Condom, oral contraceptives, etc.) are allowed to participate.

Exclusion Criteria:

* active diarrhea;
* pregnancy; breastfeeding
* 3 diarrheic episodes within 24 hours in the 15 days preceding the date of the departure;
* antibiotic treatment during the last 15 days or ongoing treatment at the time of departure;
* consumption of fermented milk, yogourt or probiotics probiotics in the 15 days preceding the date of the departure;
* immunosuppressed state or any health condition being susceptible to decompensate during the study (including malignant hemo-pathologies, AIDS, bone marrow transplant or organ transplant).
* active radiotherapy or chemotherapy as cancer treatment
* the administration of an ETEC/cholera vaccine or any other diarrhea vaccine in the three months prior to study initiation
* an active, non-controlled intestinal disease;
* ileostomy, jejunostomy or colostomy
* concomitant participation in another clinical trial
* mental or other conditions, or language barriers rendering the subject unable to understand the nature, scope, and possible consequences of the study or complete the self-administered questionnaires;
* subject unlikely to comply with protocol, e.g., uncooperative attitude, and unlikelihood of completing the study,
* allergies to any ingredients in the study product (active product or placebo)
* current use of illicit drug and alcohol abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 277 (Actual)
Dates: Start 2008-04; Primary Completion 2009-12 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
To determine the efficacy of Bio-K+ CL1285 RX® in reducing traveler's diarrhea by comparing the incidence of diarrhea in travelers during their stay abroad and upon their return to Canada, following either BIO-K+CL1285 RX® or placebo prophylaxis. | March 2008 to April 2009

SECONDARY OUTCOMES:
To compare the severity of diarrhea in travelers during their stay abroad and upon their return to Canada, following either BIO-K+CL1285 RX® or placebo prophylaxis. | March 2008 to April 2009
To compare the safety profile of BIO-K+CL1285 RX® to that of placebo | March 2008 to April 2009
To compare the physician and traveler satisfaction following daily prophylaxis with either BIO-K+CL1285 RX® or placebo | March 08 to April 09
To evaluate and compare the health economic impact of daily prophylaxis with BIO-K+CL1285 RX®. | March 08 to April 09

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Tessier, MD, Principal Investigator — Sante Voyage Medisys; Benoit Brizard, MD, Principal Investigator — Clinique Santé Voyage de Laval; Benoit Cote, MD, Principal Investigator — Clinique Sante Voyage des Prairies; Jean Vincelette, MD, Principal Investigator — Sante Voyage Saint-Luc
Locations (4):
- Canada (4):
  - Clinique Santé Voyage des Prairies, Joliette, Quebec
  - Clinique Santé Voyage de Laval, Laval, Quebec
  - Clinique Santé Voyage Saint-Luc, Montreal, Quebec
  - Sant Voyage Medisys, Montreal, Quebec